CLINICAL TRIAL: NCT03676621
Title: Buccal Misoprostol Versus IV Oxytocin in Prevention of Postpartum Hemorrhage :a Randomized Controlled Study
Brief Title: Buccal Misoprostol Versus IV Oxytocin in Prevention of Postpartum Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abo bakr mitwally, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BMISO
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patients will receive buccal misoprostol
  Interventions: Drug: Misoprostol
- control group (Active Comparator): patients will receive intravenous oxytocin
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — buccal tablets
  Arms: study group
Drug: Oxytocin — intravenous drip
  Arms: control group

SUMMARY:
Cesarean delivery is defined as fetal birth through incisions in the abdominal wall and the uterine wall (hysterotomy). This definition does not include removal of the fetus from the abdominal cavity in the case of uterine rupture or in the case of an abdominal pregnancy

DETAILED DESCRIPTION:
patients and methods:

Type of Study

A prospective registered, double blinded, randomized controlled trial

Settings and localizations:

Operative list and emergency unit at Obstetrics and Gynecology Department, Women Health Hospital, Assiut university, Egypt

Preliminary assessment of the patient

Obtain a detailed history from the patient

* Examination of the patient

  1. General examination and evaluation of the vital signs ofthe patient ( pulse , blood pressure , temperature and respiratory rate)
  2. Obstetrical examination

     Ultrasonograghic assessment (fetal viability , number of gestation, placental location, amniotic fluid index)

     Investigations ( complete blood count, Prothrombin time and concentration).

     Inclusion criteria:

     All legally adult pregnant women , above 18 years old ,at term with singleton pregnancies booked for elective caesarean section accepting to participate in the study.

     Indications of cesarean section:

     Repeated caesarean section(previous 2 cs or more).

     previous one caesarean with oligohydramnios.

     previous one caesarean with contracted pelvis.

     previous one caesarean with malpresentation.

     previous one caesarean section with decreased fetal movement.

     primigravida with malpresentation.

     primigravida with contracted pelvis.

     Exclusion criteria:

     Medical disorders involving the heart,liver,kidney or brain.

     Diabetes mellitus and hypertension.

     Patients requiring blood transfusion due to anemia.

     Risk factors for uterine atony e.g. macrosomia , polyhydramnios ,multiple pregnancies.

     Placenta previa or placental abruption.

     Previous major obstetric haemorrhage (>1000ml in previous Deliveries).

     Known fibroid or adenomyosis.

     Severe preeclampsia.

     Uterine anomalies.

     Women who received anticoagulant therapy.

     Blood disorders (e.g. coagulopathies , thrombocytopenia).

     Consent

     Verbal and written consent were obtained from all eligible women .

     The candidate women were divided into two groups. A computer generated random numerical table was used by an independent statistician to prepare sealed opaque envelopes containing a group assignment. Two groups of envelopes, corresponding to two study groups, were given to a third party (a nurse), who was unaware of the contents. The nurse distributed envelopes to patients, alternating between the groups. Patientsassigned to group 1 received 5 IU oxytocin IV after delivery of the fetus+ 2 tabs placepo . Patients assigned to group 2 received 400 in the buccal space after anaesthesia + Iv saline infusion

     Procedure:

     Cesarean deliveries were performed by well- trained resident doctor supervised by Assistant lecturer or Obstetrician consultant.

     Cesarean section was performed under spinal anesthesia. Novasoconstrictor was used unless the blood pressure dropped by 20% fromthe baseline value; if this was the case, 10 mg ephedrine was given.

     Cesarean Delivery technique was the same in all recruited women.

     Abdominal skin incision was done through a Pfannenstiel incision 2 to 3cm above the symphysis pubis, with the mid portion of the incision within the shaved area of the pubic hair for a length of about 10-12cm was done. After the rectus fascia was opened, the rectus

     muscles were separated and dissected off the peritoneum which was

     picked up between two tissue forceps and opened longitudinally. The visceral peritoneum was dissected sharply and gently to separate the bladder from the uterus. The

     uterus was opened through a transverse lower segment incision.

     After clamping of the umbilical cord, the women received 1.5 gm Ampicillin -Sulbactam (Ultracillin, Sedico, Egypt) and 80 mg garamycin (Epigent, EPICO, EGYPT)

     Uterine repair by absorbable continuous vicryl 1 sutures in two layers , parietal peritoneum was sutured by absorbable continuous vicryl sutures, rectus sheath was closed by absorbable continuous vicryl 1.

     subcutaneous fatty layer was closed by absorbable continuous vicryl 0sutures, skin was closed by vicryl 2-0 by subcuticular sutures.

     All the towels were weighed before and after cesarean section and the difference were calculated, the amount of intraoperative blood loss was estimated in the suction apparatus in ml. A trained nurse was responsible for blood and amniotic fluid collection during surgery using two separate suction sets, as well as for weighing the surgical towels before and after surgery; all towels that were used were of the same size and weight and every 1 gm increase in weight was equated with 1-mLblood loss. The total amount of intra-operative blood loss was calculated.(blood loss in suction apparatus plus weight difference of used towels

     Second trained nurse was responsible for post-operative external blood loss measurement during the first 24 hours after surgery by weighing the soaked towels placed in the vulvar area. The post-operative blood loss was calculated (weight difference of towels placed in the vulvar area .The overall blood loss was calculated. Another blood picture was obtained 24 hours postoperative to detect changes in Hb level. The same nurse was responsible for follow up body temperature 2 hours after caesarean section (feverish if temperature is 38ºC or greater) and observation of the patient for nausea , vomiting , chills and diarrhea.

     Outcomes:

     Primary outcomes: involved estimation of intraoperative and

     postoperative blood loss for 24 hours ( blood loss estimation started immediately following the skin incision)

     Secondary outcomes:

     Changes in hemoglobin concentration ( hemoglobin concentrations were measured 2 hours before surgery and 24 hours after surgery)

     Misoprostol-induced maternal adverse effects (postoperativenausea, vomiting, diarrhea, fever and chills .

     Need to use other uterotonic drugs (oxytocin or ergometrine).Need to do further surgical interventions ( uterine artery ligation ,hysterectomy or re-exploration of the patient)

     Need for blood transfusion.

     Sample Size:

     Sample size was calculated based on the primary outcome (the amount of intraoperative blood loss during cs ) based on the results of previous study ,the mean blood loss with the use of Iv oxytocinas588.9ml with a standerd deviation of 96.3 ml (10).

     Assuming that buccal misoprostol is more effective in reducing blood loss by 10% 77 participants in each group will have 95% power at significance to detect such a 5% difference

     women were include in each group taking in account a 10% 77 drop-out rate (Epi-info: centers for disease control and prevention

     Atlanta, GA)

     Approval of Ethical Considerations:

     The Research Ethics Committee of Faculty of Medicine, Assiut

     University approved the study protocol. Pregnant women who would

     undergo elective lower segment cesarean section at term ( ≥ 37 weeks)

     with normal fetal heart tracing received written and verbal information

     about the study and were asked to participate. Those who agreed signed

     an informed consent form

     Statistical Analysis:

     Data entry and analysis were carried out using Statistical Package

     of Social Sciences for windows (SPSS, Chicago, Illinois, USA) version 20

     Quantitative variables were presented in terms of mean± standard

     deviation and qualitative variables were expressed as frequency and

     percentage. Tests of significance (T-test and chi-square) were calculated

     Significance level was set at P value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* term pregnancy
* singleton pregnancies
* booked for elective cesarean section

Exclusion Criteria:

* • Medical disorders involving the heart,liver,kidney or brain

  * Diabetes mellitus and hypertension
  * Blood disorders (e.g. coagulopathies , thrombocytopenia )
  * Patients requiring blood transfusion due to anemia
  * Risk factors for uterine atony e.g. macrosomia , polyhydramnios ,multiple pregnancies
  * Placenta previa or placental abruption
  * Previous major obstetric haemorrhage (>1000ml)in previous deliveries
  * Known fibroid or adenomyosis
  * Severe preeclampsia
  * Uterine anomalies
  * Women who received anticoagulant therapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
mean blood loss | 1 hour
  the amount of blood in towels and suction drain

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt